CLINICAL TRIAL: NCT00805480
Title: Phase II Randomized, Double-blind, Multi-center, Parallel-group, Placebo-controlled Multiple-loading Dose Regimen Study to Assess the Safety, Efficacy and Duration of Response of AIN457 in Patients With Chronic Plaque-type Psoriasis.
Brief Title: Multiple-loading Dose Regimen Study in Patients With Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2212
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Plaque; psoriasis; inflammatory skin disease; skin condition, thickening; flaking; scaly patches; skin disease
MeSH Terms: conditions — Plaque, Amyloid; Psoriasis; Dermatitis; Skin Diseases | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AIN457 3 mg/kg (Experimental): Participants randomized to this arm received AIN457 3 mg/kg on day 1, and then matching placebo on days 15 and 29.
  Interventions: Drug: AIN457; Drug: Placebo
- AIN457 10 mg/kg (Experimental): Participants randomized to this arm received AIN457 10 mg/kg on day 1, and then matching placebo on days 15 and 29.
  Interventions: Drug: AIN457; Drug: Placebo
- AIN457 10 mg/kg x3 (Experimental): Participants randomized to this arm received AIN457 3 mg/kg on days 1, 15 and 29.
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator): Participants randomized to this arm received matching placebo to AIN457 on days 1, 15 and 29
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457 — AIN457 was administered intravenously.
  Other Names: Secukinumab
  Arms: AIN457 10 mg/kg; AIN457 10 mg/kg x3; AIN457 3 mg/kg
Drug: Placebo — Matching placebo to AIN457 was administered intravenously.
  Arms: AIN457 10 mg/kg; AIN457 3 mg/kg; Placebo

SUMMARY:
Loading dose, four arm, double-blind, parallel group, placebo-controlled study comparing single and multiple doses of AIN457 to placebo in patients with a diagnosis of moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis for at least 6 months prior to screening. The patients must meet all of the following criterion:

  1. Coverage of the body surface area (BSA) of 10% or more with plaques
  2. A score of 3 or more on the IGA scale
  3. A PASI score of at least 12 at baseline

     Exclusion Criteria:
* Have forms of psoriasis other than the required "plaque psoriasis"
* Women of childbearing potential
* Recent use of investigational drugs or treatment with other biological therapies (wash-out periods required)
* Previous treatment with this investigational drug
* Subjects with active or history of clinically significant cardiac, kidney or liver abnormalities;

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Novartis Investigator Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned enrollment was for 100 participants. However, one center was prematurely terminated and the data from this center could not be used for analysis. Therefore, additional participants were randomized to replace the 30 participants from the early terminated center. As a result, a total of 130 participants were enrolled.
Period: Overall Study
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Started | 30 | 29 | 31 | 10
Pharmacodynamic Analysis Set | 30 | 25 | 29 | 10
Completed | 16 | 22 | 19 | 5
Not Completed | 14 | 7 | 12 | 5
Not completed — Withdrawal by Subject | 13 | 5 | 11 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 31 | 10 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (9.29) | 43.5 (11.75) | 43.4 (10.90) | 40.1 (14.89) | 43.8 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 2 | 20
  Male | 24 | 22 | 26 | 8 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: Baseline, Week 12
Population: Participants from the PD Analysis Set, who had both baseline and week 12 values, were included in the analysis. As such, the population for each treatment group is different from the PD population in the participant flow. The PD analysis set included participants who had at least one dose of study medication and had no protocol deviations.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Number analyzed (Participants) | 27 | 23 | 27 | 5
scores on a scale | -12.46 (7.668) | -13.35 (6.195) | -18.02 (6.792) | -4.18 (4.698)

2. Primary Outcome: Percentage of Participants Who Had Not Relapsed at Any Time in the Trial
Description: This outcome measure shows the proportion of participants in each of the AIN457 treatment groups who were relapse free throughout the study up to and including week 56.
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56
Population: PD analysis set participants (AIN457 groups only), who had not yet relapsed were included in the analysis at each time point. As a result, the number of participants at risk for relapse may decrease as the number of weeks on study increases. The PD set included participants who had at least one dose of study medication and no protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3
Number analyzed (Participants) | 30 | 25 | 29
Percentage of participants
  Week 1 (n=30,25,29) | 100.0 | 100.0 | 100.0
  Week 2 (n=30,25,28) | 100.0 | 100.0 | 96.6
  Week 4 (n=30,25,27) | 100.0 | 100.0 | 93.1
  Week 6 (n=30,24,27) | 100.0 | 96.0 | 93.1
  Week 8 (n=30,24,27) | 100.0 | 96.0 | 93.1
  Week 10 (n=28,22,27) | 93.3 | 88.0 | 93.1
  Week 12 (n=23,22,27) | 76.7 | 88.0 | 93.1
  Week 14 (n=20,20,27) | 66.7 | 80.0 | 93.1
  Week 16 (n=16,19,26) | 53.3 | 76.0 | 89.7
  Week 20 (n=15,17,26) | 50.0 | 68.0 | 89.7
  Week 24 (n=13,17,25) | 43.3 | 68.0 | 86.2
  Week 28 (n=11,12,24) | 36.7 | 48.0 | 82.8
  Week 32 (n=9,9,19) | 30.0 | 36.0 | 65.5
  Week 36 (n=7,9,17) | 23.3 | 36.0 | 58.6
  Week 40 (n=6,7,14) | 20.0 | 28.0 | 48.3
  Week 44 (n=4,7,10) | 13.3 | 28.0 | 34.5
  Week 48 (n=3,6,8) | 10.0 | 24.0 | 27.6
  Week 52 (n=3,5,5) | 10.0 | 20.0 | 17.2
  Week 56 (n=2,4,5) | 12.5 | 22.2 | 27.8

3. Secondary Outcome: Percentage of Participants With at Least 50% Improvement From Baseline in PASI
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, end of study (EOS) (up to week 56)
Population: PD analysis set: The PD analysis set included participants who had at least one dose of study medication and had no major protocol deviations which could impact the PD analysis. At weeks 28, 36, 44 and 48, only 28 of the 29 participants in the AIN457 10mg/kg X3 group had values for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Number analyzed (Participants) | 30 | 25 | 29 | 10
Percentage of participants
  Week 4 | 56.7 | 84.0 | 89.7 | 10.0
  Week 8 | 73.3 | 80.0 | 93.1 | 0.0
  Week 12 | 66.7 | 79.2 | 93.1 | 10.0
  Week 16 | 50.0 | 68.0 | 89.7 | 10.0
  Week 20 | 46.7 | 68.0 | 89.7 | 10.0
  Week 24 | 40.0 | 68.0 | 86.2 | 10.0
  Week 28 (n=30,25,28,10) | 33.3 | 48.0 | 82.1 | 10.0
  Week 32 | 30.0 | 36.0 | 65.5 | 10.0
  Week 36 (n=30,25,28,10) | 23.3 | 36.0 | 51.7 | 0.0
  Week 40 | 20.0 | 28.0 | 48.3 | 10.0
  Week 44 (n=30,25,28,10) | 13.3 | 28.0 | 32.1 | 10.0
  Week 48 (n=30,25,28,10) | 6.7 | 24.0 | 28.6 | 10.0
  Week 52 | 6.7 | 20.0 | 20.7 | 0.0
  End of study (up to week 56) | 6.7 | 16.0 | 31.0 | 20.0

4. Secondary Outcome: Percentage of Participants With at Least 75% or 90% Improvement From Baseline in PASI
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, EOS (up to week 56)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Number analyzed (Participants) | 30 | 25 | 29 | 10
Percentage of participants
  Week 4 - PASI 75 | 30.0 | 56.0 | 65.5 | 0.0
  Week 4 - PASI 90 | 3.3 | 28.0 | 48.3 | 0.0
  Week 8 - PASI 75 | 53.3 | 72.0 | 89.7 | 0.0
  Week 8 - PASI 90 | 6.7 | 44.0 | 72.4 | 0.0
  Week 12 - PASI 75 | 40.0 | 75.0 | 82.6 | 10.0
  Week 12 - PASI 90 | 10.0 | 54.2 | 75.9 | 0.0
  Week 16 - PASI 75 | 30.0 | 60.0 | 82.8 | 0.0
  Week 16 - PASI 90 | 3.3 | 40.0 | 79.3 | 0.0
  Week 20 - PASI 75 | 23.3 | 52.0 | 82.8 | 0.0
  Week 20 - PASI 90 | 0.0 | 28.0 | 65.5 | 0.0
  Week 24 - PASI 75 | 20.0 | 40.0 | 69.0 | 0.0
  Week 24 - PASI 90 | 0.0 | 24.0 | 62.1 | 0.0
  Week 28 - PASI 75 (n=30,25,28,10) | 16.7 | 36.0 | 60.7 | 0.0
  Week 28 - PASI 90 (n=30,25,28,10) | 0.0 | 16.0 | 42.9 | 0.0
  Week 32 - PASI 75 | 3.3 | 24.0 | 44.8 | 0.0
  Week 32 - PASI 90 | 0.0 | 16.0 | 31.0 | 0.0
  Week 36 - PASI 75 (n=30,25,28,10) | 0.0 | 24.0 | 28.6 | 0.0
  Week 36 - PASI 90 (n=30,25,28,10) | 0.0 | 8.0 | 14.3 | 0.0
  Week 40 - PASI 75 | 0.0 | 16.0 | 21.4 | 0.0
  Week 40 - PASI 90 | 0.0 | 12.0 | 6.9 | 0.0
  Week 44 - PASI 75 (n=30,25,28,10) | 0.0 | 16.0 | 10.7 | 0.0
  Week 44 - PASI 90 (n=30,25,28,10) | 0.0 | 8.0 | 3.6 | 0.0
  Week 48 - PASI 75 (n=30,25,28,10) | 0.0 | 12.0 | 10.7 | 0.0
  Week 48 - PASI 90 (n=30,25,28,10) | 0.0 | 4.0 | 3.6 | 0.0
  Week 52 - PASI 75 | 0.0 | 12.0 | 6.9 | 0.0
  Week 52 - PASI 90 | 0.0 | 4.0 | 3.4 | 0.0
  End of study (up to week 56) - PASI 75 | 0.0 | 12.0 | 13.8 | 0.0
  End of study (up to week 56) - PASI 90 | 0.0 | 0.0 | 10.3 | 0.0

5. Secondary Outcome: Percentage of Participants in Each Investigator Global Assessment (IGA) Category
Description: The IGA scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe and 5 = very severe.
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, EOS (up to week 56)
Population: PD analysis set participants, who had values at each week category, were included in the analysis. As such, the population at each week varies from the PD population in the participant flow. The PD analysis set included participants who had at least one dose of study medication and had no major protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Number analyzed (Participants) | 30 | 25 | 29 | 10
Percentage of participants
  Baseline - Clear (n=30,25,29,10) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline - Almost clear (n=30,25,29,10) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline - Mild disease (n=30,25,29,10) | 0.0 | 0.0 | 3.4 | 0.0
  Baseline - Moderate disease (n=30,25,29,10) | 60.0 | 68.0 | 55.2 | 70.0
  Baseline - Severe disease (n=30,25,29,10) | 36.7 | 32.0 | 41.4 | 10.0
  Baseline - Very severe (n=30,25,29,10) | 3.3 | 0.0 | 0.0 | 20.0
  Week 1 - Clear (n=30,25,29,10) | 0.0 | 0.0 | 0.0 | 0.0
  Week 1 - Almost clear (n=30,25,29,10) | 3.3 | 12.0 | 13.8 | 0.0
  Week 1 - Mild disease (n=30,25,29,10) | 23.3 | 32.0 | 48.3 | 10.0
  Week 1 - Moderate disease (n=30,25,29,10) | 66.7 | 56.0 | 37.9 | 70.0
  Week 1 - Severe disease (n=30,25,29,10) | 6.7 | 0.0 | 0.0 | 10.0
  Week 1 - Very severe disease (n=30,25,29,10) | 0.0 | 0.0 | 0.0 | 10.0
  Week 2 - Clear (n=30,25,27,10) | 0.0 | 4.0 | 6.9 | 0.0
  Week 2 - Almost clear (n=30,25,27,10) | 3.3 | 20.0 | 24.1 | 10.0
  Week 2 - Mild disease (n=30,25,27,10) | 50.0 | 64.0 | 44.8 | 0.0
  Week 2 - Moderate disease (n=30,25,27,10) | 46.7 | 12.0 | 17.2 | 80.0
  Week 2 - Severe disease (n=30,25,27,10) | 0.0 | 0.0 | 0.0 | 0.0
  Week 2 - Very severe disease (n=30,25,27,10) | 0.0 | 0.0 | 0.0 | 10.0
  Week 4 - Clear (n=30,25,27,9) | 0.0 | 16.0 | 17.2 | 0.0
  Week 4 - Almost clear (n=30,25,27,9) | 16.7 | 32.0 | 44.8 | 0.0
  Week 4 - Mild disease (n=30,25,27,9) | 46.7 | 44.0 | 24.1 | 20.0
  Week 4 - Moderate disease (n=30,25,27,9) | 36.7 | 8.0 | 6.9 | 40.0
  Week 4 - Severe disease(n=30,25,27,9) | 0.0 | 0.0 | 0.0 | 20.0
  Week 4 - Very severe disease (n=30,25,27,9) | 0.0 | 0.0 | 0.0 | 10.0
  Week 6 - Clear (n=30,24,27,7) | 0.0 | 24.0 | 31.0 | 0.0
  Week 6 - Almost clear (n=30,24,27,7) | 23.3 | 28.0 | 48.3 | 0.0
  Week 6 - Mild disease (n=30,24,27,7) | 50.0 | 32.0 | 10.3 | 0.0
  Week 6 - Moderate disease (n=30,24,27,7) | 26.7 | 12.0 | 3.4 | 60.0
  Week 6 - Severe disease(n=30,24,27,7) | 0.0 | 0.0 | 0.0 | 0.0
  Week 6 - Very severe disease(n=30,24,27,7) | 0.0 | 0.0 | 0.0 | 10.0
  Week 8 - Clear (n=30,24,27,7) | 0.0 | 28.0 | 41.4 | 0.0
  Week 8 - Almost clear (n=30,24,27,7) | 33.3 | 32.0 | 34.5 | 0.0
  Week 8- Mild disease (n=30,24,27,7) | 40.0 | 20.0 | 13.8 | 0.0
  Week 8 - Moderate disease(n=30,24,27,7) | 26.7 | 16.0 | 3.4 | 60.0
  Week 8 - Severe disease (n=30,24,27,7) | 0.0 | 0.0 | 0.0 | 0.0
  Week 8 - Very severe disease (n=30,24,27,7) | 0.0 | 0.0 | 0.0 | 10.0
  Week 10 - Clear (n=28,24,25,5) | 0.0 | 28.0 | 48.3 | 0.0
  Week 10 - Almost clear (n=28,24,25,5) | 30.0 | 28.0 | 31.0 | 0.0
  Week 10 - Mild disease (n=28,24,25,5) | 36.7 | 20.0 | 6.9 | 0.0
  Week 10 - Moderate disease (n=28,24,25,5) | 26.7 | 16.0 | 0.0 | 40.0
  Week 10 - Severe disease (n=28,24,25,5) | 0.0 | 4.0 | 0.0 | 10.0
  Week 10 - Very severe disease (n=28,24,25,5) | 0.0 | 0.0 | 0.0 | 0.0
  Week 12 - Clear (n=27,23,27,5) | 0.0 | 32.0 | 48.3 | 0.0
  Week 12 - Almost clear (n=27,23,27,5) | 26.7 | 16.0 | 27.6 | 0.0
  Week 12 - Mild disease (n=27,23,27,5) | 33.3 | 16.0 | 13.8 | 10.0
  Week 12- Moderate disease (n=27,23,27,5) | 16.7 | 20.0 | 3.4 | 30.0
  Week 12 - Severe disease (n=27,23,27,5) | 13.3 | 8.0 | 0.0 | 10.0
  Week 12 - Very severe disease (n=27,23,27,5) | 0.0 | 0.0 | 0.0 | 0.0
  Week 14 - Clear (n=22,22,26,4) | 0.0 | 32.0 | 58.6 | 0.0
  Week 14 - Almost clear (n=22,22,26,4) | 16.7 | 12.0 | 17.2 | 0.0
  Week 14 - Mild disease (n=22,22,26,4) | 30.0 | 24.0 | 10.3 | 0.0
  Week 14 - Moderate disease (n=22,22,26,4) | 16.7 | 8.0 | 3.4 | 30.0
  Week 14 - Severe (n=22,22,26,4) | 10.0 | 12.0 | 0.0 | 10.0
  Week 14 - Very severe (n=22,22,26,4) | 0.0 | 0.0 | 0.0 | 0.0
  Week 16 - Clear (n=20,21,26,4) | 0.0 | 24.0 | 55.2 | 0.0
  Week 16 - Almost clear(n=20,21,26,4) | 13.3 | 24.0 | 20.7 | 0.0
  Week 16 - Mild disease(n=20,21,26,4) | 23.3 | 16.0 | 10.3 | 10.0
  Week 16 - Moderate disease (n=20,21,26,4) | 20.0 | 12.0 | 3.4 | 10.0
  Week 16 - Severe disease (n=20,21,26,4) | 6.7 | 8.0 | 0.0 | 20.0
  Week 16 - Very severe disease (n=20,21,26,4) | 3.3 | 0.0 | 0.0 | 0.0
  Week 20 - Clear (n=17,18,26,3) | 0.0 | 12.0 | 44.8 | 0.0
  Week 20 - Almost clear (n=17,18,26,3) | 6.7 | 32.0 | 20.7 | 10.0
  Week 20 - Mild disease (n=17,18,26,3) | 33.3 | 8.0 | 20.7 | 0.0
  Week 20 - Moderate disease (n=17,18,26,3) | 10.0 | 20.0 | 3.4 | 20.0
  Week 20 - Severe disease (n=17,18,26,3) | 6.7 | 0.0 | 0.0 | 0.0
  Week 20 - Very severe disease (n=17,18,26,3) | 0.0 | 0.0 | 0.0 | 0.0
  Week 24 - Clear (n=15,18,26,3) | 0.0 | 8.0 | 37.9 | 0.0
  Week 24 - Almost clear (n=15,18,26,3) | 6.7 | 28.0 | 31.0 | 10.0
  Week 24 - Mild disease(n=15,18,26,3) | 30.0 | 12.0 | 10.3 | 0.0
  Week 24 - Moderate disease(n=15,18,26,3) | 10.0 | 20.0 | 10.3 | 20.0
  Week 24 - Severe disease(n=15,18,26,3) | 3.3 | 4.0 | 0.0 | 0.0
  Week 24 - Very severe disease(n=15,18,26,3) | 0.0 | 0.0 | 0.0 | 0.0
  Week 28 - Clear (n=14,17,24,2) | 0.0 | 4.0 | 13.8 | 0.0
  Week 28 - Almost clear (n=14,17,24,2) | 3.3 | 28.0 | 24.1 | 10.0
  Week 28 - Mild disease (n=14,17,24,2) | 23.3 | 4.0 | 37.9 | 0.0
  Week 28 - Moderate disease (n=14,17,24,2) | 16.7 | 24.0 | 6.9 | 10.0
  Week 28 - Severe disease (n=14,17,24,2) | 3.3 | 8.0 | 0.0 | 0.0
  Week 28 - Very severe disease (n=14,17,24,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 32 - Clear (n=11,12,23,2) | 0.0 | 8.0 | 10.3 | 0.0
  Week 32 - Almost clear (n=11,12,23,2) | 0.0 | 12.0 | 24.1 | 0.0
  Week 32 - Mild disease (n=11,12,23,2) | 20.0 | 16.0 | 27.6 | 10.0
  Week 32 - Moderate disease (n=11,12,23,2) | 16.7 | 8.0 | 13.8 | 10.0
  Week 32 - Severe disease (n=11,12,23,2) | 0.0 | 4.0 | 3.4 | 0.0
  Week 32 - Very severe disease (n=11,12,23,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 36 - Clear (n=9,9,19,2) | 0.0 | 4.0 | 6.9 | 0.0
  Week 36 - Almost clear (n=9,9,19,2) | 0.0 | 12.0 | 13.8 | 0.0
  Week 36 - Mild disease (n=9,9,19,2) | 16.7 | 8.0 | 20.7 | 0.0
  Week 36 - Moderate disease (n=9,9,19,2) | 13.3 | 12.0 | 20.7 | 20.0
  Week 36 - Severe disease (n=9,9,19,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 36 - Very severe disease (n=9,9,19,2) | 0.0 | 0.0 | 3.4 | 0.0
  Week 40 - Clear (n=8,8,18,2) | 0.0 | 8.0 | 3.4 | 0.0
  Week 40 - Almost clear (n=8,8,18,2) | 0.0 | 8.0 | 10.3 | 0.0
  Week 40 - Mild disease (n=8,8,18,2) | 6.7 | 4.0 | 31.0 | 0.0
  Week 40 - Moderate disease (n=8,8,18,2) | 20.0 | 12.0 | 17.2 | 20.0
  Week 40 - Severe disease (n=8,8,18,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 40 - Very severe disease (n=8,8,18,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 44 - Clear (n=6,8,14,2) | 0.0 | 0.0 | 3.4 | 0.0
  Week 44 - Almost clear (n=6,8,14,2) | 0.0 | 12.0 | 3.4 | 0.0
  Week 44 - Mild disease (n=6,8,14,2) | 6.7 | 4.0 | 13.8 | 10.0
  Week 44 - Moderate disease (n=6,8,14,2) | 13.3 | 16.0 | 20.7 | 10.0
  Week 44 - Severe disease (n=6,8,14,2) | 0.0 | 0.0 | 6.9 | 0.0
  Week 44 - Very severe disease (n=6,8,14,2) | 0.0 | 0.0 | 0.0 | 0.0
  Week 48 - Clear (n=3,7,11,1) | 0.0 | 0.0 | 3.4 | 0.0
  Week 48 - Almost clear (n=3,7,11,1) | 0.0 | 8.0 | 0.0 | 0.0
  Week 48 - Mild disease (n=3,7,11,1) | 3.3 | 8.0 | 17.2 | 0.0
  Week 48 - Moderate disease (n=3,7,11,1) | 6.7 | 12.0 | 17.2 | 10.0
  Week 48 - Severe disease (n=3,7,11,1) | 0.0 | 0.0 | 0.0 | 0.0
  Week 48 - Very severe disease (n=3,7,11,1) | 0.0 | 0.0 | 0.0 | 0.0
  Week 52 - Clear (n=3,7,10,0) | 0.0 | 0.0 | 3.4 | 0.0
  Week 52 - Almost clear (n=3,7,10,0) | 0.0 | 8.0 | 0.0 | 0.0
  Week 52 - Mild disease (n=3,7,10,0) | 6.7 | 4.0 | 6.9 | 0.0
  Week 52 - Moderate disease (n=3,7,10,0) | 3.3 | 16.0 | 17.2 | 0.0
  Week 52 - Severe disease (n=3,7,10,0) | 0.0 | 0.0 | 6.9 | 0.0
  Week 52 - Very severe disease (n=3,7,10,0) | 0.0 | 0.0 | 0.0 | 0.0
  End of study - Clear (n=12,8,13,5) | 0.0 | 0.0 | 6.9 | 0.0
  End of study - Almost clear (n=12,8,13,5) | 3.3 | 4.0 | 3.4 | 0.0
  End of study - Mild disease (n=12,8,13,5) | 6.7 | 8.0 | 3.4 | 20.0
  End of study - Moderate disease (n=12,8,13,5) | 30.0 | 16.0 | 27.6 | 30.0
  End of study - Severe disease (n=12,8,13,5) | 0.0 | 4.0 | 3.4 | 0.0
  End of study - Very severe disease (n=12,8,13,5) | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | AIN457 3 mg/kg | AIN457 10 mg/kg | AIN457 10 mg/kg x3 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/30 | 3/29 | 2/31 | 0/10
Other Adverse Events (participants affected / at risk) | 15/30 | 22/29 | 19/31 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 3 mg/kg (N=30) | AIN457 10 mg/kg (N=29) | AIN457 10 mg/kg x3 (N=31) | Placebo (N=10)
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 1 | 0
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 | 0 | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 3 mg/kg (N=30) | AIN457 10 mg/kg (N=29) | AIN457 10 mg/kg x3 (N=31) | Placebo (N=10)
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 2 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 4 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 9 | 8 | 4 | 0
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1 | 2 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 5 | 3 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
BLOOD AMYLASE INCREASED (Investigations) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 2 | 5 | 0
DEPRESSION (Psychiatric disorders) | 0 | 3 | 0 | 0
HYPERTENSION (Vascular disorders) | 4 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.